CLINICAL TRIAL: NCT02805088
Title: Interaction Emotion-cognition in the Study of Literal and Figurative Language in Schizophrenia and Bipolar Disorders: Behavioral and Electrophysiological Studies
Brief Title: Emotions in Schizophrenia and Bipolar Disorders: a Common Vulnerability?
Acronym: ELISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: PO13116
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Bipolar Disorder; Schizophrenia
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia

ARMS (3):
- Bipolar Disorder patients (Experimental)
  Interventions: Other: Electroencephalographic recordings; Other: neuropsychological evaluation; Other: clinical evaluation of symptoms
- Schizophrenia patients (Experimental)
  Interventions: Other: Electroencephalographic recordings; Other: neuropsychological evaluation; Other: clinical evaluation of symptoms
- Healthy Volunteers (Experimental)
  Interventions: Other: Electroencephalographic recordings; Other: neuropsychological evaluation; Other: clinical evaluation of symptoms

INTERVENTIONS:
Other: Electroencephalographic recordings
Other: neuropsychological evaluation
Other: clinical evaluation of symptoms

SUMMARY:
The initial aim of the project was to gain an understanding of the comprehension of "language-oriented" emotions among schizophrenic and bipolar patients. By "language-oriented" emotions, the investigators mean the emotions that are conveyed by means of language, whether through the emotional valence of the words, the expression of an emotional state or emotional prosody. Although they involve different diagnostic categories, schizophrenic and bipolar disorders nevertheless share a number of symptoms, in particular in the emotional sphere, and do so to such an extent that the question of whether there may, at the clinical, cognitive and etiopathogenic levels, exist a continuum between these disorders is frequently raised. Taking this hypothesis of a clinical continuum as our starting point, the investigators explored the understanding of emotions contextualized by language in these two clinical populations, namely patients exhibiting schizophrenic and bipolar disorders. To these populations, the investigators also added the dimension of vulnerability in the form of non-clinical participants varying in terms of their traits of schizotypy and hypomania, thus orienting this project toward the early identification of cognitive-emotional markers and possibly also their prevention.

DETAILED DESCRIPTION:
The aim of this proposal is to investigate disturbances of understanding of "emotional language" in schizophrenia and bipolar disorder. By "emotional langague", the investigators mean emotions wich can be drawn from utterances, thanks to affective valence of words or phrases, expression of emotional state or prosody. Schizophrenia and bipolar disorder share several symptoms, particularly those related to emotional sphere, in such a way that it is frequently asked whether these disorders could be formalized on a continuum. Comparing the cognitive-emotional functioning of these two kinds of patients should allow identifying cognitive markers of the psychotic symptom dimension common in both diseases.

On the basis of the abundant literature regarding cognitive-emotional functioning in schizophrenia and on the more infrequent literature concerning bipolar functioning, the investigators hypothesized that the difficulties in processing emotions, in attributing intentionality and in integrating information for meaning are markers for the psychotic symptom dimension common in both pathologies. To test this hypothesis, the investigators chose to investigate language understanding because it can imply a semantic-emotional processing and because it necessitates integration processes. The integration processes obligatory operate on semantic information, from which it can be added, in ecological situations, prosodic and intentional information. The proposed methodology involves different levels of language, requiring more or less complex integration processes - literal language and figurative language - and different emotional features - affective valence of words and expressions and emotional prosody -.

The investigators plan to conduct behavioral and electrophysiological (event-related potentials) studies. For the later, The investigators will focus on electrophysiological components well known to be implied in language and emotional processing: the N400, the LPC (Late Positive Component) and the LPP (Late Positive Potential). The combination of behavioral and electrophysiological indicators will allow the identification of the neurocognitive mechanisms shared by both schizophrenic and bipolar patients, particularly those who experienced a psychotic episode, in comparison with those of healthy participants. These studies will be conducted on 60 stable schizophrenic patients, 60 euthymic bipolar patients with or without psychotic symptoms, and 120 healthy participants, matched on age and educational achievement level to each pathological group. Different instruments will be used to investigate, in both pathological groups and their controls, different emotional dimensions (anhedonia, alexithymia, positive or negative affectivity, depression, anxiety). Investigating the cognitive-emotional functioning of patients from a dimensional approach (psychotic symptom dimension) rather than from a categorical approach could impulse a new way of thinking diagnosis or identifying factors of vulnerability and protection for these diseases.

ELIGIBILITY:
Inclusion criteria

Patients :

Men or women, right-handed, with a diagnosis of bipolar disorder or schizophrenia, according to the DSM-IV criteria, aged from 18 to 65 years-old Native French speaker Clinically stabilised Able to provide informed written and verbal consent

Healthy Controls :

Men or women, right-handed, aged from 18 to 65 years-old Native French speaker Able to provide informed written and verbal consent

Exclusion criteria

Patients :

A recent alcohol and/or drug abuse or dependence A significant general medical illness, including neurological disorders or head trauma A sensorial impairment (visual and/or hearing)

Healthy Controls :

A personal or first-degree-relative history of bipolar disorder, schizophrenia or schizoaffective disorder according to DSM-IV A recent alcohol and/or drug abuse or dependence A significant general medical illness, including neurological disorders or head trauma A sensorial impairment (visual and/or hearing)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Event-related brain potentials (ERP) | within 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France

REFERENCES:
- [Result] Terrien S, Gobin P, Iakimova G, Coutte A, Thuaire F, Baltazart V, Mazzola-Pomietto P, Besche-Richard C. Electrophysiological correlates of emotional meaning in context in relation to facets of schizotypal personality traits: A dimensional study. Psychiatry Clin Neurosci. 2016 Mar;70(3):141-50. doi: 10.1111/pcn.12366. Epub 2015 Dec 22. PMID 26482112
- [Result] Terrien S, Gobin P, Coutte A, Thuaire F, Iakimova G, Mazzola-Pomietto P, Besche-Richard C. Emotional Meaning in Context in Relation to Hypomanic Personality Traits: An ERP Study. PLoS One. 2015 Sep 22;10(9):e0138877. doi: 10.1371/journal.pone.0138877. eCollection 2015. PMID 26394230
- [Result] Terrien S, Stefaniak N, Morvan Y, Besche-Richard C. Factor structure of the French version of the Hypomanic Personality Scale (HPS) in non-clinical young adults. Compr Psychiatry. 2015 Oct;62:105-13. doi: 10.1016/j.comppsych.2015.07.001. Epub 2015 Jul 8. PMID 26343474